CLINICAL TRIAL: NCT03851146
Title: A Phase I Investigation of the Safety, Tolerability and Immunological Effects of T Lymphocytes Transduced With an Anti-Lewis Y (LeY) Chimeric Antigen Receptor Gene (LeY-CAR-T) in Patients With LeY Antigen Expressing Advanced Solid Tumours
Brief Title: A Study of Anti-Lewis Y Chimeric Antigen Receptor-T Cells (LeY-CAR-T) in Patients With Solid Tumours
Acronym: LeY-CAR-T
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LeYPh1-02; ACTRN12616001580460 (Other: ANZCTR)
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Intervention Model Description: The study will employ dose level cohorts of three patients that will be treated at each level described in Table 1, based on the number of T cells to be infused using the "3 + 3" dose-escalation strategy. If the proposed number of T cells is unable to be obtained due to technical production reasons, the available number will be infused. However, the cohort will only be escalated when a minimum of three patients have been safely treated at the planned level.
  The fourth cohort dose level has been set according to the maximum level considered to be feasible taking into account technical constraints. The study will be expanded to accrue additional patients at the MTD (expansion phase cohort) with an expansion cohort of upto 20 patients. For technical and logistic reasons the maximum number of patients to be enrolled on the study will be 30.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LeY CAR T cells (Experimental): One arm study consisting of "3 + 3" dose escalation study design (see below) followed by dose expansion phase at determined MTD.
  Dose level : Target Number LeY CART cells infused *
  -1 (if needed): 1 x 10e8
  1. 2 x 10e8
  2. 5 x 10e8
  3. 1 x 10e9
  4. 5 x 10e9
     * Targeted number of LeY CAR T cells (minus 40% acceptance range) for manufacture according toTGA-approved standard protocols
  Treatment follows a lymphodepleting, chemotherapy regimen that consists of Fludarabine (25 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) for 3 consecutive days prior to cell infusion, with chemotherapy completed at least 48 hours before the re-infusion of the LeY CAR T cells.
  Interventions: Biological: LeY CAR T cells

INTERVENTIONS:
Biological: LeY CAR T cells — Autologous peripheral blood T-lymphocytes transduced with the anti-LeY-scFv-CD28-ζ vector (LeY CAR T cells)

SUMMARY:
This clinical trial is an open-label, single-centre, phase I study designed to investigate the safety and tolerability of a single infusion of autologous peripheral blood T-lymphocytes transduced with the anti-LeY-scFv-CD28-ζ vector (LeY CAR T-cells) The primary aim of the trial is to evaluate the safety and tolerability of LeY CAR T cells in patients with Lewis Y antigen-expressing, advanced solid tumours.

The secondary aim of the trial is to assess the anti-tumour activity of LeY CAR T cells in patients with LeY antigen-expressing, advanced solid tumours.

Patients aged 18 years or older with advanced solid tumours have consented to pre-screening that allows their tumours to be assessed for LeY expression by immunohistochemistry. Patients whose tumours test positive for LeY were then able to proceed to eligibility screening and, if found to fulfil the eligibility criteria, were registered in the study. The study involves an initial dose escalation phase followed by an expansion phase.

DETAILED DESCRIPTION:
To autologous peripheral blood T-lymphocytes transduced with the anti-LeY-scFv-CD28-ζ vector in patients with LeY expressing advanced solid tumours. evaluate the safety and tolerability of an intravenous infusion of autologous peripheral blood T-lymphocytes transduced with the anti-LeY-scFv-CD28-ζ vector in patients with LeY expressing advanced solid tumours.

Aims:

To evaluate the safety and tolerability of an intravenous infusion of autologous peripheral blood T-lymphocytes transduced with the anti-LeY-scFv-CD28-ζ vector in patients with LeY expressing advanced solid tumours.

Primary Objectives To determine the maximum tolerated dose and rate of dose limiting toxicities of a single intravenous infusion of autologous peripheral blood T-lymphocytes transduced with the anti-LeY-scFv-CD28-ζ vector in patients with LeY expressing advanced solid tumours (LeY CAR T cells).

Secondary Objectives i. To assess the anti-tumour activity of the LeY CAR T cells in terms of overall response, duration of response, progression free survival and overall survival.

ii. To assess persistence in peripheral blood of the LeY CAR T cells.

The study will recruit an anticipated number of 12 patients in the dose escalation phase consisting of 4 dose levels, each with dose level cohorts of 3 patients. Following completion of the dose-escalation phase, additional patients with Le Y expressing solid tumours will be recruited to the study. These patients will be administered the maximum number of cells safely delivered in the dose escalation phase of the study. A subset comprising 5 patients in the expansion cohort will be administered Indium-111 labelled T-cells and imaged by SPECT to determine the biodistribution of reinfused T cells.

If the proposed number of T cells is unable to be obtained due to technical production reasons, the available number will be infused.

It is anticipated that up to 30 patients will be treated on this protocol.

ELIGIBILITY:
Inclusion Criteria:

All of the following must apply at the time of enrollment:

1. Patients with an advanced solid tumour (defined as incurable locally advanced or metastatic disease and excluding any haematologic malignancy).

   Tumour is positive for Lewis Y expression by immunohistochemistry - defined as a staining of ≥ 10 % of tumour cells positive for LeY expression. For the purposes of tumour screening, where possible the most recently available tumour sample should be utilised. A new biopsy is not mandatory where archival tissue is available, but may be considered.
2. Patient is ≥18 years of age.
3. Patient has an ECOG performance status of 0 - 1
4. Patient has provided written confirmation of informed consent on participant information and consent form
5. Life expectancy of ≥ 12 weeks
6. Patient has adequate organ function satisfying all of the following:

   * Liver: bilirubin <1.5x upper limit of normal (ULN) unless patient has known Gilbert's syndrome;
   * AST/ALT ≤2.5 x ULN except in patients with known liver metastases where AST/ALT≤5.0
   * Kidney: either serum creatinine <1.5x ULN or creatinine clearance > 50ml/min. Creatinine clearance is either derived using the Cockcroft-Gault formula or may be measured by 24 hour urine collection or nuclear medicine assessment.
   * Lung: Adequate pulmonary function defined by SaO2 >91% on room air and ≤ grade I dyspnoea.
   * Cardiac: LVEF ≥ 40% as confirmed by echocardiogram or multiple uptake gated acquisition (MUGA)
   * Adequate bone marrow reserve as defined as:

     * Absolute neutrophil count (ANC) ≥ 1.0 x 10e9/L
     * Absolute lymphocyte count ≥ 0.5 x 10e9/L
     * Platelets ≥ 100 x 10e9/L
     * Haemoglobin >80g/L
     * WCC <30 x 10e9/L
7. Patient is deemed capable and willing to undergo the planned study procedures in the view of the principal investigator.
8. Women of childbearing potential (defined as all women physiologically capable of becoming pregnant) and all male participants must agree to use highly effective methods of contraception for one year following LeY CART therapy.
9. Patient has measurable disease as per RECIST 1.1.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in this study:

1. Patients with known active central nervous system (CNS) involvement by malignancy. Patients with previous treated and/or neurologically stable disease will be eligible.
2. Prior chimeric antigen receptor T (CART) cell therapy
3. Patient has been given chemotherapy and/or G-CSF in the last 4 weeks or is planned to receive such therapy prior to apheresis of PBMC. Patients can only receive cytotoxic drugs as per the schedule of treatment for this protocol.
4. Patient has had immunosuppressive therapy within 4 weeks of apheresis. Therapeutic doses of steroids (defined as > 20 mg/day of Prednisolone (or equivalent) must be able to be stopped > 7 days prior to leukapheresis and 72 hours prior to LeY CART cell infusion Physiologic doses of steroid (e.g. Prednisolone <10mg or equivalent), topical and inhaled steroids are permitted.
5. Patient who are eligible for potentially curative therapy
6. Uncontrolled active or latent Hepatitis B or active Hepatitis C or HIV
7. Patients with uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics.
8. History or presence of active clinically relevant CNS pathology such as epilepsy, aphasia, severe brain injury, dementia, Parkinson's disease, cerebellar disease or psychosis.
9. Radiation therapy within 2 weeks prior to registration
10. Patient has an active haematologic malignancy (any lymphoma, leukaemia, multiple myeloma or myelodysplastic syndrome)
11. Patient has a history of significant pulmonary disease (including radiation pneumonitis) or known, biopsy proven autoimmune inflammatory disease of the gastrointestinal tract.
12. Unstable angina or myocardial infarct within 6 months prior to screening.
13. Patient has known clinically significant autoimmune disease with positive serology for RHF (>20kU/L) or ANA (titre >1:40).
14. Women of child bearing potential (WOCBP) who are unwilling or unable to use an effective method of contraception to avoid pregnancy for the entire study period and for at least 12 months after completion of study treatment.
15. Women who are pregnant or breastfeeding.
16. Men who are unwilling or unable to use an acceptable method of contraception for the entire study period and for at least 12 months after completion of study treatment if their sexual partners are WOCBP.
17. Patient has a serious uncontrolled medical disorder, psychological or social factors that which would impair the ability to receive protocol therapy and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerated Dose (MTD) of LeY CAR T-cell infusion | 4 weeks
  To determine the maximum tolerated dose of a single intravenous infusion of Le Y CAR T-cells in patients with LeY expressing advanced solid tumours.This outcome will be assessed by evaluating occurrence, type, severity and relationship to treatment of adverse events (AEs) according to NCI CTCAE v4.03 and laboratory abnormalities.
  To be reported as Total Number of Le Y CAR T-cells infused eg. Y x 10e(9)
The Dose-Limiting Toxicities (DLTs) associated with LeY CAR T-cell infusion | 4 weeks
  To determine the rate of dose limiting toxicities of a single intravenous infusion of Le Y CAR T-cells in patients with LeY expressing advanced solid tumours.
  DLT Definition:
  1. Any treatment-emergent Grade 4 or 5 (death) AEs related to LeY CAR T cells, excluding laboratory values deemed not clinically significant.
  2. Any treatment-emergent Grade 3 AEs related to LeY CAR T cells that do not resolve to ≤ Grade 2 within 7 days, excluding laboratory values deemed not clinically significant
  3. Any treatment-emergent Grade 3 or 4 seizure
  4. Any treatment-emergent autoimmune event ≥ Grade 3.
  All Adverse Events(AEs) will recorded in the eCRF using the severity grade according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

SECONDARY OUTCOMES:
To assess the Overall Response (OR) to anti-tumour activity of LeY CAR T-cells | 5 years
  Overall response (OR), defined as the best response to the CAR T-cells re-infusion based on RECIST v1.1 criteria. Response will be determined by CT scan at baseline (screening), week 4 and week 8 post-infusion, every 8 weeks thereafter until 1 year has elapsed, followed by every 12 weeks until progression.
  The main analysis will occur once all patients have had 12 months follow up with the final analysis to occur once all patients have had 5 years follow-up.
To assess the Duration of Response (PR) to anti-tumour activity of LeY CAR T-cells | 5 years
  Duration of response, defined as the time from the date of first response of PR or better until the date of disease progression, for those patients who experience a PR or better as assessed by RECIST v1.1 criteria (death is a censoring event), for those patients who experience a PR or better.
  Response will be determined by CT scan at baseline (screening), week 4 and week 8 post-infusion, every 8 weeks thereafter until 1 year has elapsed, followed by every 12 weeks until progression.
  The main analysis will occur once all patients have had 12 months follow up with the final analysis to occur once all patients have had 5 years follow-up.
To assess the Progression Free Survival (PFS) of patients treated with LeY CAR T-cells | 5 years
  Progression free survival (PFS), defined as the time from LeY CAR T cells re-infusion to the earliest of date of disease progression as assessed by RECIST v1.1criteria or death.
  Response will be determined by CT scan at baseline (screening), week 4 and week 8 post-infusion, every 8 weeks thereafter until 1 year has elapsed, followed by every 12 weeks until progression.
  The main analysis will occur once all patients have had 12 months follow up with the final analysis to occur once all patients have had 5 years follow-up.
To assess the Overall Survival (OS) of patients treated with LeY CAR T-cells | 5 years
  Overall survival (OS), defined as the time from LeY CAR T cells re-infusion to date of death.
  Response will be determined by CT scan at baseline (screening), week 4 and week 8 post-infusion, every 8 weeks thereafter until 1 year has elapsed, followed by every 12 weeks until progression.
  The main analysis will occur once all patients have had 12 months follow up with the final analysis to occur once all patients have had 5 years follow-up.
To assess persistence of anti-LeY T-cells in peripheral blood | 12 months
  Detection (presence/absence) and quantification of LeY CAR T-cell transgene in peripheral blood by qPCR at each of the following time points of assessment (day -7(pre-infusion), day 0 (day of infusion), days 1, 2, 3, 6, 10, 14, 21, 28, 42, 56 post-infusion and every 4 weeks thereafter until 1 year has elapsed.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Solomon, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyran D, Zhu JJ, Butler J, Tantalo D, MacDonald S, Nguyen TN, Wang M, Thio N, D'Souza C, Qin VM, Slaney C, Harrison A, Sek K, Petrone P, Thia K, Giuffrida L, Scott AM, Terry RL, Tran B, Desai J, Prince HM, Harrison SJ, Beavis PA, Kershaw MH, Solomon B, Ekert PG, Trapani JA, Darcy PK, Neeson PJ. TSTEM-like CAR-T cells exhibit improved persistence and tumor control compared with conventional CAR-T cells in preclinical models. Sci Transl Med. 2023 Apr 5;15(690):eabk1900. doi: 10.1126/scitranslmed.abk1900. Epub 2023 Apr 5. PMID 37018415